CLINICAL TRIAL: NCT04831723
Title: NEWBIE Validate: Feasibility of a New Test to Measure Glucose in Newborn Blood Spots (NBS)
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2107147
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Neonatal Diabetes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this feasibility laboratory study is to evaluate whether the laboratory testing pathway for glucose screening in newborn blood spots (NBS) can be done at scale, and that the glucose test has a carefully established cut-off to define what level glucose is abnormal at day 5 of life.

The investigators aim to run this feasibility study for a period of 6 to 12 months to fully embed and test the process. This will equate to assessing glucose levels in approximately 10,000 NBS samples. The results from this study will inform a future large scale prospective screening study.

ELIGIBILITY:
Inclusion Criteria:

* Babies having a routine NBS screening test.
* Routine maternity care team within the area served by the Portsmouth regional screening laboratory (NHS Trusts within Hampshire, Dorset & parts of Wiltshire)

Exclusion Criteria:

* Parent decides to opt-out of the blood glucose test feasibility study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Babies having a routine NBS screening test within the areas served by the Portsmouth regional screening laboratory (NHS Trusts within Hampshire, Dorset & parts of Wiltshire)
Sampling Method: Non-Probability Sample
Enrollment: 10784 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Normal range of capillary blood glucose in newborns at day 5 of life | 12 months

SECONDARY OUTCOMES:
Validation of laboratory procedures | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Mcdonald, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Dorset County Hospital, Dorchester
  - University Hospitals Dorset, Poole
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No